CLINICAL TRIAL: NCT01130103
Title: Combination Treatment for PTSD After the WTC Attack
Brief Title: Combination Treatment for Posttraumatic Stress Disorder (PTSD) After the World Trade Center (WTC) Attack
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Franklin Schneier, Research Psychiatrist, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH068173 (NIH); R01MH068173 (NIH)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; anxiety disorders; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Wounds and Injuries | interventions — Paroxetine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxetine (Experimental): Paroxetine and Prolonged Exposure Therapy
  Interventions: Drug: Paroxetine; Behavioral: Prolonged Exposure Therapy
- Placebo pill (Placebo Comparator): Placebo pill plus Prolonged Exposure Therapy
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Drug: Paroxetine — Paroxetine (controlled release) 12.5-50 milligrams (mg) daily for 22 weeks
  Other Names: Paxil controlled release (CR)
  Arms: Paroxetine
Behavioral: Prolonged Exposure Therapy — Weekly for 10 weeks
  Other Names: Cognitive Behavioral Therapy

SUMMARY:
This randomized controlled trial evaluates efficacy of combined prolonged exposure (PE) and the selective serotonin reuptake inhibitor (SSRI) paroxetine in the treatment of survivors of the World Trade Center (WTC) attacks.

DETAILED DESCRIPTION:
Selective serotonin reuptake inhibitor (SSRI) medication is often recommended in combination with cognitive behavioral therapies for PTSD, but combined initial treatment of PTSD has not been studied under controlled conditions. Also, there are few studies of either treatment in survivors of terrorism. This randomized controlled trial evaluates efficacy of combined prolonged exposure (PE) and the SSRI paroxetine in the treatment of survivors of the World Trade Center (WTC) attacks.

ELIGIBILITY:
Inclusion Criteria:

* Posttraumatic Stress Disorder, chronic, related to World Trade Center Attacks
* Age 18-70
* CAPS score greater than 45
* Willingness to consent
* For women, negative pregnancy test and using adequate birth control

Exclusion Criteria:

* Prominent suicidal ideation
* Current psychotic disorder
* Unstable medical illness
* Women who are pregnant or nursing mothers
* Alcohol or substance use disorder in the past 3 months
* History of seizure disorder
* conditions that contraindicate use of paroxetine
* inability to tolerate a drug free period prior to beginning the study of 4 weeks for MAOIs or fluoxetine and 2 weeks for other psychotropic drugs, except zolpidem for insomnia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Schneier FR, Neria Y, Pavlicova M, Hembree E, Suh EJ, Amsel L, Marshall RD. Combined prolonged exposure therapy and paroxetine for PTSD related to the World Trade Center attack: a randomized controlled trial. Am J Psychiatry. 2012 Jan;169(1):80-8. doi: 10.1176/appi.ajp.2011.11020321. Epub 2011 Sep 9. PMID 21908494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: December, 2004 to February, 2009. Location: Anxiety Disorders research clinic.
Period: Randomized Treatment
Arm/Group | Paroxetine | Placebo Pill
Started | 19 | 18
Completed | 13 | 13
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Maintenance Treatment
Arm/Group | Paroxetine | Placebo Pill
Started | 13 | 13
Completed | 11 | 11
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine | Placebo Pill | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: PTSD severity, minimum = 0 = no symptoms of PTSD maximum = 136 = extremely severe symptoms of PTSD
Time Frame: Weeks 0,5,10
Population: all participants who were randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo Pill
Number analyzed (Participants) | 19 | 18
units on a scale
  week 0 | 72.6 (12.9) | 65.4 (12.8)
  week 5 | 40.7 (28.4) | 49.0 (23.9)
  week 10 | 21.5 (19.9) | 35.6 (31.3)
Statistical Analysis 1: Comparison: Paroxetine vs Placebo Pill; caps total score at weeks 5 and 10; Test type: Superiority or Other; p = .01, Mixed Models Analysis; incident rate ratio = 0.50, 95% CI 2-sided [.30 to .85]
Statistical Analysis 2: Comparison: Paroxetine vs Placebo Pill; rate of change in CAPS total from week 5 to week 10; Test type: Superiority or Other; p < .001, Mixed Models Analysis; incident rate ratio = .56, 95% CI 2-sided [.43 to .74]

2. Secondary Outcome: Treatment Response at Weeks 5 and 10
Description: responder status: CGI-change score of 1 or 2
  1=very much improved, 2= much improved
Time Frame: weeks 5,10
Population: all subjects randomized with dropouts carried forward as nonresponders
Measure: Number; unit: participants
Arm/Group | Paroxetine | Placebo Pill
Number analyzed (Participants) | 19 | 18
participants
  week 5 | 6 | 6
  week 10 | 12 | 7

3. Secondary Outcome: Hamilton Depression Scale 0 = no Depression Symptoms 40 = Extreme Depression Symptoms
Description: total score at weeks 0, 5, 10
Time Frame: weeks 0,5,10
Population: observed data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo Pill
Number analyzed (Participants) | 19 | 18
units on a scale
  week 0 | 16.9 (4.9) | 16.6 (4.9)
  week 5 | 11.7 (5.9) | 11.8 (5.6)
  week 10 | 7.7 (3.7) | 11.4 (6.7)

4. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Scale Total Score at Week 0,5,10
Description: Measures life enjoyment and satisfaction across 16 domains 16 = very poor quality of life to 80 =very good quality of life
Time Frame: weeks 0,5,10
Population: observed data at weeks 0, 5, and 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo Pill
Number analyzed (Participants) | 16 | 16
units on a scale
  week 0 | 47.1 (11.0) | 45.4 (18.5)
  week 5 | 55.5 (13.4) | 59.4 (17.6)
  week 10 | 67.9 (12.7) | 54.8 (22.3)

5. Primary Outcome: Number of Participants Who Met Remission Criterion
Description: remission defined as: CAPS less than or equal to 20 and Clinical Global Impression (CGI)-change score=1
Time Frame: Weeks 5,10
Population: all participants who were randomized, with people who dropped out counted as non-remitters
Measure: Number; unit: participants
Arm/Group | Paroxetine | Placebo Pill
Number analyzed (Participants) | 19 | 18
participants
  week 5 | 2 | 0
  week 10 | 8 | 3
Statistical Analysis 1: Comparison: Paroxetine vs Placebo Pill; treatment group effect: remission rate at weeks 5 and 10; Test type: Superiority or Other; p = .03, Mixed Models Analysis; Odds Ratio (OR) = 12.6, 95% CI 2-sided [1.23 to 129]
Statistical Analysis 2: Comparison: Paroxetine vs Placebo Pill; rate of change over time in remission rate from week 5 to 10; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; Odds Ratio (OR) = 20.8, 95% CI 2-sided [2.44 to 176]

ADVERSE EVENTS:
Arm/Group | Paroxetine | Placebo Pill
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 6/19 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine (N=19) | Placebo Pill (N=18)
headache (Nervous system disorders) | 2 (2) | 2 (2)
palpitations (Cardiac disorders) | 2 (2) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
sweating (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
photophobia (Eye disorders) | 2 (2) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
constipation (Gastrointestinal disorders) | 4 (4) | 2 (2)
diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2)
lightheadedness (Nervous system disorders) | 1 (1) | 3 (3)
dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
blurry vision (Eye disorders) | 3 (3) | 1 (1)
parasthesias (Nervous system disorders) | 1 (1) | 3 (3)
decrease libido (Reproductive system and breast disorders) | 4 (4) | 0 (0)
anorgasmia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
impaired coordination (Nervous system disorders) | 3 (3) | 2 (2)
nervousness (Nervous system disorders) | 3 (3) | 1 (1)
fatigue (General disorders) | 3 (3) | 3 (3)
insomnia (Nervous system disorders) | 1 (1) | 2 (2)
weight gain (General disorders) | 2 (2) | 1 (1)
weight loss (General disorders) | 2 (2) | 3 (3)
skin problems (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
difficulty urinating (Renal and urinary disorders) | 2 (2) | 4 (4)
rigidity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
somnolence (General disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No